CLINICAL TRIAL: NCT03291769
Title: Effects of Intraoperative Blood Transfusion on Postoperative Results in Pediatric Cardiac Surgery
Brief Title: Effects of Intraoperative Blood and Blood Product Consumption on Postoperative Results in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Specialist doctor, Cukurova University
Other Study IDs: PHS01
Record Dates: First submitted 2017-08-23; First posted 2017-09-25 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Blood Loss, Surgical; Pediatric Heart Surgery
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood products and intravenous fluids are frequently used in the treatment of children who have undergone cardiac surgery in order to maintain hemodynamic stability. Optimal hematocrit values during CPB are still being discussed in children undergoing congenital cardiac surgery. The overall complication rate for transfusion in adults is 2.5 complications per 1000 units, while 10.7 complications per 1000 transfusion in children. The aim of this study is to investigate the effects of the our transfusion strategies used in pediatric cardiac surgery on duration of intensive care unit, duration of postoperative mechanical ventilation and mortality.

DETAILED DESCRIPTION:
Background: Blood products and intravenous fluids are frequently used in the treatment of children who have undergone cardiac surgery in order to maintain hemodynamic stability. Children undergoing cardiac surgery with cardiopulmonary bypass (CPB) are among the greatest pediatric users of allogeneic red blood cells (RBCs), and transfusions are used in 79% of all procedures. Optimal hematocrit values during CPB are still being discussed in children undergoing congenital cardiac surgery. While it is argued that high hematocrit values provide better results in perioperative period and postoperative neurological development, it is also argued that blood products are associated with mortality and morbidity. The overall complication rate for transfusion in adults is 2.5 complications per 1000 units, while 10.7 complications per 1000 transfusion in children.

Balancing the benefits and risks of blood transfusion is a particularly complex issue, especially in children. Because many aspects of transfusion therapy in children are not well researched.

Method: This prospective, observational study will be conducted following Cukurova University Faculty of Medicine Ethics Committee approval. Children aged 16 years or younger who will undergo open heart surgery due to congenital heart disease will be included in the study. Patients with preoperative renal or hepatic disease will be excluded. Age, comorbidities, history of previous operation will be recorded. Preoperative hematocrit, biochemical parameters (blood urea nitrogen, creatinine, electrolytes), cardiac profile (angiography and echocardiography reports, diagnosis of the disease requiring the surgery) and preoperative medications, preoperative RACHS1 (risk adjustment for congenital heart disease, risk management for congenital heart disease) will be recorded.

In the intraoperative period; the haematocrit values before CPB, during CPB, after CPB and after reversal of the heparin with protamine will be recorded. Aortic cross clamp time, body temperature, urine volume and diuretic use during CPB will be recorded. Blood gas values, central venous oxygen saturation (SvO2) and lactate levels will be recorded in the intraoperative period within 30 min intervals. The amount of crystalloid and colloid, erythrocyte, fresh frozen plasma, platelet and cryoprecipitate used in the intraoperative period will be recorded. The ACT (active coagulation time) values at the beginning and at the end of the operation, the amount of applied heparin and protamine will be recorded. Vasoactive agents (dopamine, dobutamine, adrenaline, nitroglycerin) used in the intraoperative period will be recorded.

In the postoperative intensive care unit; blood gas and lactate values, hematocrit, chest tube drainage and iv fluids (crystalloid and colloid) and blood products will be recorded at postoperative 6th and 24th hours. The vasoactive agents, the inotrope score, the amount of urine and the use of diuretics will be recorded. The length of stay in intensive care unit, the duration of mechanical ventilation will be recorded.

Major complications will be identified as cardiac arrest, neurological deficit (stroke, seizure), acute renal failure requiring dialysis therapy, arrhythmia requiring permanent heart pace and multiple organ dysfunction and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 16 years or younger who will undergo heart surgery due to congenital heart disease will be included in the study.

Exclusion Criteria:

* Children with renal failure
* Children with hepatic disease

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child
Study Population: Children aged 16 years or younger who will undergo heart surgery due to congenital heart disease will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Length of stay in intensive care unit | Postoperative 3 months
  Postoperative length of stay in intensive care unit

SECONDARY OUTCOMES:
Mortality | Postoperative 3 months
  Postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Feri̇de Karacaer, Study Director — Cukurova University
Locations (1):
- Feri̇de Karacaer, Adana, In the USA Or Canada, Please Select..., Turkey (Türkiye)

REFERENCES:
- [Background] Rizza A, Romagnoli S, Ricci Z. Fluid Status Assessment and Management During the Perioperative Phase in Pediatric Cardiac Surgery Patients. J Cardiothorac Vasc Anesth. 2016 Aug;30(4):1085-93. doi: 10.1053/j.jvca.2015.11.007. Epub 2015 Nov 10. No abstract available. PMID 26944520